CLINICAL TRIAL: NCT00078858
Title: Prolonged Mycophenolate Mofetil and Truncated Cyclosporine Postgrafting Immunosuppression to Reduce Life-Threatening GVHD After Unrelated Donor Peripheral Blood Cell Transplantation Using Nonmyeloablative Conditioning for Patients With Hematologic Malignancies and Renal Cell Carcinoma - A Multi-Center Trial
Brief Title: Mycophenolate Mofetil and Cyclosporine in Reducing Graft-Versus-Host Disease in Patients With Hematologic Malignancies or Metastatic Kidney Cancer Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1668.00; NCI-2012-00668 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1668.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA018029 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2019-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Childhood Renal Cell Carcinoma; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Clear Cell Renal Cell Carcinoma; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Juvenile Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Renal Cell Cancer; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Anemia; Refractory Anemia With Ringed Sideroblasts; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Splenic Marginal Zone Lymphoma; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Childhood Anaplastic Large Cell Lymphoma; Stage I Childhood Large Cell Lymphoma; Stage I Childhood Lymphoblastic Lymphoma; Stage I Childhood Small Noncleaved Cell Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Childhood Anaplastic Large Cell Lymphoma; Stage II Childhood Large Cell Lymphoma; Stage II Childhood Lymphoblastic Lymphoma; Stage II Childhood Small Noncleaved Cell Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Childhood Anaplastic Large Cell Lymphoma; Stage III Childhood Large Cell Lymphoma; Stage III Childhood Lymphoblastic Lymphoma; Stage III Childhood Small Noncleaved Cell Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Childhood Anaplastic Large Cell Lymphoma; Stage IV Childhood Large Cell Lymphoma; Stage IV Childhood Lymphoblastic Lymphoma; Stage IV Childhood Small Noncleaved Cell Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Renal Cell Cancer; T-cell Large Granular Lymphocyte Leukemia; Type 1 Papillary Renal Cell Carcinoma; Type 2 Papillary Renal Cell Carcinoma; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Carcinoma, Renal Cell; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Anemia, Refractory; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (prolonged MMF and truncated CSP) (Experimental): CONDITIONING: Patients receive fludarabine phosphate IV over 30 minutes on days -4 to -2, and undergo TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBMC transplant on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO BID on days -3 to 80 with taper to day 150 and mycophenolate mofetil PO or IV TID on days 0-30, BID on days 31-150, and then taper to day 180. Treatment continues in the absence of unacceptable toxicity.
  Interventions: Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBMC transplantation
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic PBMC transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: cyclosporine — Given PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies whether stopping cyclosporine before mycophenolate mofetil is better at reducing the risk of life-threatening graft-versus-host disease (GVHD) than the previous approach where mycophenolate mofetil was stopped before cyclosporine. The other reason this study is being done because at the present time there are no curative therapies known outside of stem cell transplantation for these types of cancer. Because of age or underlying health status, patients may have a higher likelihood of experiencing harm from a conventional blood stem cell transplant. This study tests whether this new blood stem cell transplant method can be made safer by changing the order and length of time that immune suppressing drugs are given after transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the incidence of life-threatening GVHD can be reduced after unrelated donor peripheral blood mononuclear cell (PBMC) hematopoietic cell transplantation (HCT) using nonmyeloablative conditioning with earlier discontinuation of cyclosporine (CSP) and extended administration of mycophenolate mofetil (MMF) in patients with hematologic malignancies and metastatic renal cell carcinoma.

SECONDARY OBJECTIVES:

I. To compare the incidence of acute and chronic GVHD to protocols 1463 and 1641.

II. To compare the utilization of corticosteroids to protocols 1463 and 1641.

III. To compare survival to that achieved under protocol 1463 and 1641.

OUTLINE:

CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -4 to -2, and undergo total-body irradiation (TBI) on day 0.

TRANSPLANTATION: Patients undergo allogeneic PBMC transplant on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) twice daily (BID) on days -3 to 80 with taper to day 150 and mycophenolate mofetil PO or IV thrice daily (TID) on days 0-30, BID on days 31-150, and then taper to day 180. Treatment continues in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 24 months and then yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 50 years with hematologic malignancies treatable by unrelated HCT
* Ages =< 50 years of age with hematologic diseases treatable by allogeneic HCT who through pre-existing medical conditions or prior therapy are considered to be at high risk for regimen related toxicity associated with a conventional transplant (> 40% risk of transplant-related mortality [TRM]) or those patients who refuse a conventional HCT; transplants must be approved for these inclusion criteria by both the participating institution's patient review committee such as the Patient Care Conference (PCC at the Fred Hutchinson Cancer Research Center [FHCRC]) and by the principal investigator at the collaborating center; patients =< 50 years of age who have received previous high-dose transplantation do not require patient review committee approval; all children < 12 years must be discussed with the FHCRC primary investigator (PI) prior to registration
* Patients with metastatic renal cell carcinoma with the histologic subtypes of clear cell, papillary and medullary may be accepted regardless of age
* The following diseases will be permitted although other diagnoses can be considered if approved by PCC or the participating institution's patient review committees and the principal investigator:

  * Aggressive non-Hodgkin lymphomas (NHLs) and other histologies such as diffuse large B cell NHL-not eligible for autologous hematopoietic stem cell transplant (HSCT), not eligible for conventional myeloablative HSCT, or after failed autologous HSCT
  * Low grade NHL- with < 6 month duration of complete remission (CR) between courses of conventional therapy
  * Mantle cell NHL-may be treated in first CR
  * Chronic lymphocytic leukemia (CLL)- Must be refractory to fludarabine; patients who fail to have a complete or partial response after therapy with a regimen containing fludarabine (or another nucleoside analog, e.g. 2-cladribine [CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing fludarabine (or another nucleoside analog)
  * Hodgkin disease (HD)- must have received and failed frontline therapy
  * Multiple myeloma (MM)- must have received prior chemotherapy; consolidation of chemotherapy by autografting prior to nonmyeloablative HCT is permitted
  * Acute myeloid leukemia (AML)- must have < 5% marrow blasts at the time of transplant.
  * Acute lymphocytic leukemia (ALL)- must have < 5% marrow blasts at the time of transplant
  * Chronic myelogenous leukemia (CML)- Patients will be accepted in chronic phase or accelerated phase; patients who have received prior autografts after high dose therapy or have undergone intensive chemotherapy with filgrastim (G-CSF)-mobilized peripheral blood mononuclear cells (G-PBMC) autologous or conventional HCT for advanced CML may be enrolled provided they are in CR or CP and have < 5% marrow blasts at time of transplant
  * Myelodysplastic syndrome (MDS)/myeloproliferative disorder (MPD)- Only patients with MDS/refractory anemia (RA) or MDS/refractory anemia with ringed sideroblasts (RARS) will be eligible for this protocol; additionally patients with myeloproliferative syndromes (MPS) will be eligible; those patients with MDS or MPS with > 5% marrow blasts (including those with transformation to AML) must receive cytotoxic chemotherapy and achieve < 5% marrow blasts at time of transplant
  * Renal cell carcinoma- Must have evidence of disease not amenable to surgical cure or history of or active metastatic disease by radiological and histologic criteria
* DONOR: FHCRC matching allowed will be grade 1.0 to 2.1: Unrelated donors who are prospectively:

  * Matched for human leukocyte antigen (HLA)-A, B, C, major histocompatibility complex, class II, DR beta 1 (DRB1) and major histocompatibility complex, class II, DQ beta 1 (DQB1) by high resolution typing;
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* DONOR: A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
* DONOR: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0201, and this type of mismatch is not allowed
* DONOR: G-PBMC only will be permitted as a HSC source on this protocol

Exclusion Criteria:

* Patients with rapidly progressive intermediate or high grade NHL
* Renal cell carcinoma patients

  * With expected survival of less than 6 months
  * Disease resulting in severely limited performance status (< 70%)
  * Any vertebral instability
  * History of brain metastases
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant
* Patients with non-hematological tumors except renal cell carcinoma
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Cardiac ejection fraction < 35%; ejection fraction is required if there is a history of anthracycline exposure or history of cardiac disease
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 40% and/or receiving supplementary continuous oxygen
* The FHCRC PI of the study must approve of enrollment of all patients with pulmonary nodules
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bridging fibrosis, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease
* Karnofsky scores < 60 (except renal cell carcinoma [RCC])
* Patients with > grade II hypertension by Common Toxicity Criteria (CTC)
* Human immunodeficiency virus (HIV) positive patients
* The addition of cytotoxic agents for "cytoreduction" with the exception of hydroxyurea and imatinib mesylate will not be allowed within two weeks of the initiation of conditioning
* DONOR: Marrow donors
* DONOR: Donors who are HIV-positive and/or, medical conditions that would result in increased risk for G-CSF mobilization and harvest of G-PBMC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-09; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Incidence of life-threatening GVHD in patients undergoing a modified taper of post-grafting immunosuppression after undergoing nonmyeloablative HSCT from matched unrelated donors | 1 year
  Life-threatening GVHD defined as (1) death related to GVHD or its treatment, (2) disability caused by GVHD or its treatment (3) 3 or more major infections in a calendar year or (4) suicidal ideation because of GVHD.

SECONDARY OUTCOMES:
Need for corticosteroid treatment, defined as more than 1 mg/kg or equivalent of prednisone for more than 3 days at any time after transplant | 1 year
Graft rejection | Up to day 365
Incidence of acute and chronic GVHD | Up to 7 years
Overall survival | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (10):
- United States (7):
  - Stanford University Hospitals and Clinics, Stanford, California
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert Memorial Lutheran Hospital, Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (2):
  - Universitaet Leipzig, Leipzig
  - University of Tuebingen-Germany, Tübingen
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241